CLINICAL TRIAL: NCT05734599
Title: NMR-based Metabolic Profiling Identifies High Risk of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD) Patients With Advanced Fibrosis: An Observational, Multi-center Study
Brief Title: NMR-based Metabolic Profiling Identifies High Risk of MAFLD Patients With Advanced Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Other Study IDs: MAFLD-NMR 2022
Record Dates: First submitted 2023-01-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Dysfunction-associated Fatty Liver Disease; Metabolic Disease
Keywords: NMR-profiling; advanced fibrosis
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood and urine samples are collected from participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MAFLD-control group: Participants accepted health examinations including vibration-controlled transient elastography in Tongji and Union hospitals who are not MAFLD patients and are willing to participate in this study.
  Interventions: Device: NMR-based metabolic profiling
- MAFLD-high hardness group: Participants accepted health examinations including vibration-controlled transient elastography in Tongji and Union hospitals who are defined to have MAFLD and are willing to participate in this study.
  The risk of advanced liver fibrosis was estimated based on the LSM value, FIB-4 score, and NAFLD fibrosis score (NFS), and patients were then divided into groups of low and high hardness according to the risk measured, as shown below:
  High hardness group:
  participants meet one of the following three requirements: LSM≥ 11.4 kPa；9.9<LSM≤11.4 kPa and NFS≥0.676;9.9<LSM≤11.4 kPa and FIB-4≥2.67.
  NFS = -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m2) + 1.13 × Fasting blood glucose abnormalities / diabetes mellitus (with=1, none=0) + 0.99 × AST/ALT ratio - 0.013 × platelets (×109/L) - 0.66 × albumin (g/dl) FIB-4 = （age(years) x AST [U/L]) / ((PLT [109/L]) x (ALT [U/L])^(1/2))
  Interventions: Device: NMR-based metabolic profiling
- MAFLD-low hardness group: Participants accepted health examinations including vibration-controlled transient elastography in Tongji and Union hospitals who are defined to have MAFLD and are willing to participate in this study.
  The risk of advanced liver fibrosis was estimated based on the LSM value, FIB-4 score, and NAFLD fibrosis score (NFS), and patients were then divided into groups of low and high hardness according to the risk measured, as shown below:
  Low hardness group:
  participants who do not meet the requirements of the high hardness group are low hardness group: LSM < 9.9 kPa；9.9<LSM≤11.4 kPa with NFS < 0.676 and FIB-4<2.67.
  NFS = -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m2) + 1.13 × Fasting blood glucose abnormalities / diabetes mellitus (with=1, none=0) + 0.99 × AST/ALT ratio - 0.013 × platelets (×109/L) - 0.66 × albumin (g/dl) FIB-4 = （age(years) x AST [U/L]) / ((PLT [109/L]) x (ALT [U/L])^(1/2))
  Interventions: Device: NMR-based metabolic profiling

INTERVENTIONS:
Device: NMR-based metabolic profiling — Clinical parameters and VCTE results of each patient will be collected. Patients will be grouped into two groups according to VCTE, FIB-4 and NFS, and undergo NMR-based metabolic profiling

SUMMARY:
This study aim to find out metabolic molecules in blood and urine which could identify high risk of advanced fibrosis in MAFLD patients via NMR-based metabolic profiling.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated fatty liver disease (MAFLD) is currently the most common liver disease in the world, with an incidence of 29.81% in China. Studies have shown that the severity of liver fibrosis is the most important predictor of disease progression in patients with MAFLD, and the more severe the degree of liver fibrosis, the worse the prognosis. Therefore, discovering non-invasive indicators that can predict the risk and identify people at high risk of MAFLD with advanced liver fibrosis is essential for early clinical intervention in order to improve their clinical prognosis. Some non-invasive tests like Vibration-controlled Transient Elastography (VCTE), Fibrosis-4 Index (FIB-4), and NAFLD fibrosis score (NFS) have been used to evaluate the liver fibrosis state in MAFLD patients, but lack of prospect in metabolic molecular level. Nuclear magnetic resonance(NMR)-based metabolomic profiling can identify and quantify significant biological molecules in tissue extracts, body fluids (blood, urine, cerebrospinal fluid, saliva, etc.), and secretions, and has wide applications in the study of cancer and other metabolic diseases. Therefore, this study intends to collect the demographic characteristics and serological indicators of MAFLD patients detected by liver VCTE, and use NMR profiling to perform metabolomic analysis on their peripheral blood and urine samples, in order to discover potential non-invasive biomarkers that can be used to predict and evaluate MAFLD advanced liver fibrosis, and further verify these MAFLD metabolomic indicators that may be associated with advanced liver fibrosis through multi-center clinical studies, in an attempt to provide ideal non-invasive biomarkers for MAFLD progression prediction and clinical intervention monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MAFLD

  * Meet the diagnostic criteria in the 2020 Asian Pacific Association for the Study of the Liver (APASL) Clinical Practice Guidelines for the Diagnosis and Management of Metabolism-Related Fatty Liver Disease
  * Liver Vibration-controlled Transient Elastography (FibroTouch) with evidence of hepatic steatosis (CAP value≥ 240db/m)
  * Age≥ 18 years

Healthy controls:

* Liver Vibration-controlled Transient Elastography (FibroTouch) showed no fatty liver and no liver fibrosis;
* No history of other chronic diseases, no use of appropriate prescription drugs;
* The amount of alcohol consumed was ≤8 g per day for women and ≤16g per day for men.

Exclusion Criteria:

* • Chronic viral hepatitis, alcoholic liver disease or excessive alcohol consumption (more than 30 g of alcohol per day for men and 20 g for women), decompensated cirrhosis;

  * Chronic liver disease due to other causes (e.g., autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, hereditary hemochromatosis, Wilson disease, alpha-1 antitrypsin deficiency, celiac disease)
  * Imaging findings suggest a malignant mass of the liver;
  * Patients with other malignant tumors (excluding cured ones);
  * Have secondary obesity due to endocrine, genetic, metabolic, and central nervous system diseases. Judge by professional doctors whether it is hypothalamic obesity, pituitary obesity, hypothyroid obesity, obesity caused by Cushing's syndrome and hypogonadal obesity;
  * Have received or are currently receiving medical or surgical treatment for weight loss in the past three months or are currently being treated;
  * Weight fluctuations of ≥ 5 kg over the past two months;
  * Currently pregnant or nursing;
  * Severe cardiovascular and cerebrovascular disease or stage III hypertension;
  * Hepatitis B, active tuberculosis, AIDS and other infectious diseases;
  * Those who are unable to sign the informed consent form (such as mental illness and drug addiction, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort selected patients with and without MAFLD who underwent VCTE and serological tests.
Sampling Method: Non-Probability Sample
Enrollment: 1194 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
NMR profiling to discover the difference of lipids and lipoproteins in peripheral blood and urine that can be used to predict liver fibrosis in MAFLD progression | follow-up up to 24 months
  NMR-based metabolic profiling was used to detect and compare the lipids and lipoproteins of peripheral blood samples of control groups and MAFLD participants including the high and low hardness groups as mentioned above.
NMR profiling to discover the difference of lipoproteins in peripheral blood and urine that can be used to predict liver fibrosis in MAFLD progression | follow-up up to 24 months
  NMR-based metabolic profiling was used to detect and compare the lipoproteins of peripheral blood samples of control groups and MAFLD participants including the high and low hardness groups as mentioned above.
NMR profiling to discover the difference of amino acid and their derivatives in peripheral blood and urine that can be used to predict liver fibrosis in MAFLD progression | follow-up up to 24 months
  NMR-based metabolic profiling was used to detect and compare the amino acid and its derivatives of peripheral blood and urine samples of control groups and MAFLD participants including the high and low hardness groups as mentioned above.
NMR profiling to discover the difference of Carbohydrates and their derivatives in peripheral blood and urine that can be used to predict liver fibrosis in MAFLD progression | follow-up up to 24 months
  NMR-based metabolic profiling was used to detect and compare the Carbohydrates and their derivatives of peripheral blood and urine samples of control groups and MAFLD participants including the high and low hardness groups as mentioned above.

SECONDARY OUTCOMES:
Insulin resistance index (HOMA-IR) comparison between control groups and MAFLD participants. | follow-up up to 24 months
  The insulin resistance index in different groups, as mentioned above, were calculated and analyzed, in order to explore the factors associated with insulin resistance and diabetes in MAFLD.
  HOMA-IR=（FPG×FINS）/22.5, FPG (mmol/L), FINS(mIU/L)

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China